CLINICAL TRIAL: NCT05504590
Title: Comparison of Tuohy Needle and Quincke Needle on the Incidence of Intravascular Injection During Caudal Epidural Injection Under Ultrasound Guidance: Prospective Randomized Controlled Study
Brief Title: Comparison of Tuohy Needle and Quincke Needle During Caudal Epidural Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2022-0238
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Caudal Epidural Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuohy needle group (Experimental): Ultrasound-guided caudal epidural block with Touhy needle
  Interventions: Device: Tuohy needle group
- Quincke needle group (Active Comparator): Ultrasound-guided caudal epidural block with Quincke needle
  Interventions: Device: Quincke needle group

INTERVENTIONS:
Device: Tuohy needle group — Ultrasound-guided caudal epidural block with Touhy needle
  Arms: Tuohy needle group
Device: Quincke needle group — Ultrasound-guided caudal epidural block with Quincke needle
  Arms: Quincke needle group

SUMMARY:
Park et al. reported the results of a randomized study of the use of ultrasound and the use of C-arm in caudal epidural block. However, it is difficult to determine the overall epidural space contrast agent spread with ultrasound alone, and intravascular injection can be avoided with ultrasound. It was said that the evidence for the efficacy of exclusion of intravascular infusion was not as good as that of the C-arm. Therefore, it was suggested that ultrasound in caudal epidural block should be considered only when it is difficult to use the C-arm as an auxiliary means to guide the needle when the sacral hiatus is less than 2 mm and has a complex anatomical structure. The purpose of this study is to determine the difference between intravascular injection and epidural spread according to the type of needle during caudal block under ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

1. A patient who visited the pain clinic complaining of lower back pain due to lumbar disc/stenosis
2. When NRS of back and/or radiating pain is 4 or more
3. Patients over 19 years of age

Exclusion Criteria:

1. Malignancy
2. Systemic infection
3. Bleeding tendency
4. Contrast Allergy
5. Pregnant women
6. If you cannot read or agree to the consent form
7. If you cannot sign the consent form yourself

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
incidence of intravascular injection | 1 minute after finishing caudal epidural block
  incidence of intravascular injection during caudal epidural block

SECONDARY OUTCOMES:
time required to complete caudal epidural block | Baseline, 1 second after the completion of caudal epidural block
  time required to complete caudal epidural block

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JY, Lee JS, Kim JY, Baek JW, Kim HS, Kim DH. Comparison of the incidence of intravascular injection using the Tuohy and Quincke needles during ultrasound-guided caudal epidural block: a prospective randomized controlled study. Reg Anesth Pain Med. 2024 Jan 11;49(1):17-22. doi: 10.1136/rapm-2023-104504. PMID 37169489